CLINICAL TRIAL: NCT06507007
Title: Genetic and Epigenetic Background of Inner Ear Dysfunction in Turner Syndrome
Acronym: EPIHEAR
Status: Recruiting | Type: Observational
Sponsor: Gødstrup Hospital (Other)
Collaborators: University of Aarhus (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Louise Hill-Madsen, Medical Doctor, Gødstrup Hospital
Other Study IDs: LHM-TS-2024
Record Dates: First submitted 2024-06-24; First posted 2024-07-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Sensorineural Hearing Loss; Turner Syndrome; Inner Ear Disease
Keywords: Epigenetics; Sensorineural hearing loss; Turner Syndrome; Inner Ear Dysfunction
MeSH Terms: conditions — Hearing Loss, Sensorineural; Turner Syndrome; Labyrinth Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Individuals with TS and SNHL
- Group 2: Individuals with TS without SNHL
- Group 3: Healthy age matched controls without TS and without SNHL

SUMMARY:
The goal of this case-control study is to pave the way for new revolutionary treatment measures within hearing loss that could either replace or delay the need for hearing aids. The study focuses on people with Turner syndrome (TS).

The aim is to find out if there are specific DNA methylation patterns and/or RNA expression profiles linked to sensorineural hearing loss (SNHL) in people with TS. Additionally, the structure and function of the inner ear in these individuals will be examined to see if there is a connection to their epigenetic profile.

The main question it aims to answer is: Does epigenetics constitute a common denominator for some of the unexplained SNHL cases?

Turner Syndrome (TS) represents an ideal model for studying epigenetics related to sensorineural hearing loss (SNHL).

Participants will undergo the following tests:

* Ear examinations
* Hearing tests
* Balance tests
* Blood tests
* MRI scans
* CBCT (cone-beam computed tomography) scans

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60 years old

Exclusion Criteria:

* Contraindications for the MRI or CBCT
* Serious medical disorders
* Neurological or psychiatric disorders of any kind
* Use of medication that is known to influence inner ear function
* Medical history with dizziness or hearing problems (controls only)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Three different populations will be included as it is expected that 50% of the TS population suffer from SNHL:
  * 50 individuals with TS and SNHL
  * 50 individuals with TS without SNHL
  * 50 healthy controls without TS and SNHL
  The participants are recruited from an existing cohort.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Epigenetic profile | 2024-2026
  DNA methylation analyses are conducted on the purified DNA. RNA expression analyses and ChIP-seq are performed on the purified RNA. Based on this, the epigenetic profile will be mapped to identify consistent differences associated with SNHL.

SECONDARY OUTCOMES:
Hearing ability | 2024-2026
  Hearing level thresholds and bone conduction is assesed by pure tone audiometry.
Vestibular status | 2024-2026
  The vestibular function is assessed using the video head impulse test (vHIT), vestibular evoked myogenic potentials, and posturography.
Structural malformations | 2024-2026
  Anatomy and inner ear malformations are examined using Conebeam CT and MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Therese Ovesen, Prof, Principal Investigator — University Clinic of Flavour, Balance and Sleep
Locations (1):
- ENT department of Gødstrup Hospital, Herning, Denmark